CLINICAL TRIAL: NCT03511768
Title: A Study of 18F-AlF-NOTA-octreotide PET/CT for Imaging Neuroendocrine Neoplasms
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201801001
Record Dates: First submitted 2018-04-17; First posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Neuroendocrine Neoplasm
Keywords: 18F-AlF-NOTA-octreotide
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Al18F-NOTA-octreotide; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-AlF-NOTA-octreotide PET/CT (Experimental): One injection of the radioligand 18F-AlF-NOTA-octreotide
  Interventions: Drug: 18F-AlF-NOTA-octreotide; Device: PET/CT

INTERVENTIONS:
Drug: 18F-AlF-NOTA-octreotide — One injection of 18F-AlF-NOTA-octreotide
  Other Names: 18F-IMP466
Device: PET/CT — Following injection of 18F-AlF-NOTA-octreotide the participants will be subjected to whole body PET/CT

SUMMARY:
The aim of this study is to investigate the clinical value of [18F]aluminum fluoride-1,4,7-triazacyclononane-1,4,7-triacetic acid-octreotide（18F-AlF-NOTA-octreotide ） positron emission tomography / computed tomography (PET/CT) in patients with neuroendocrine neoplasms (NENs).

DETAILED DESCRIPTION:
18F-AlF-NOTA-octreotide is a radioligand targeting the somatostatin receptor, which is widely expressed on the cell surface of NENs. The radioligand can be used for the diagnosis and stage of the NENs. A total of 5 volunteers and 60 NEN patients will be subjected to a 18F-AlF-NOTA-octreotide PET/CT scan. The uptake of 18F-AlF-NOTA-octreotide in organs and tumor lesions will be quantified as Standardized Uptake Values (SUVmax/SUVmean).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or clinically confirmed and/or suspicious of NEN.
2. Signed informed consent.

Exclusion Criteria:

1. Claustrophobia (unable to accept PET/CT scanning)
2. Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
18F-AlF-NOTA-octreotide PET/CT imaging of patients with Neuroendocrine Neoplasms | 12 months
  The radioligand 18F-AlF-NOTA-octreotide can be used to visualize neuroendocrine neoplasms

SECONDARY OUTCOMES:
18F-AlF-NOTA-octreotide PET/CT prognostic factor for overall and disease specific survival | 24 months
  The uptake of the 18F-AlF-NOTA-octreotide in neuroendocrine neoplasm lesions (quantified as Standard Uptake Values) is associated with overall and disease specific free survival (PFS) neuroendocrine neoplasms

CONTACTS AND LOCATIONS:
Overall Officials: Tingting Long, MD,Phd, Principal Investigator — Department of PET Center,Xiangya Hospital, Central South University
Locations (1):
- Department of PET Center,Xiangya Hospital,Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Laverman P, McBride WJ, Sharkey RM, Eek A, Joosten L, Oyen WJ, Goldenberg DM, Boerman OC. A novel facile method of labeling octreotide with (18)F-fluorine. J Nucl Med. 2010 Mar;51(3):454-61. doi: 10.2967/jnumed.109.066902. Epub 2010 Feb 11. PMID 20150268